CLINICAL TRIAL: NCT05686213
Title: ExeNTrO: Exercise During Neoadjuvant Chemoradiation Treatment to Improve Rectal and
Brief Title: ExeNTrO: Exercise During Neoadjuvant Chemoradiation Treatment to Improve Rectal and Esophageal Cancer Outcome - Pilot Trial
Acronym: ExeNTrO
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NL81016.091.22
Record Dates: First submitted 2022-11-09; First posted 2023-01-17 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2022-11

CONDITIONS: Oncology
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- combined aerobic exercise + resistance exercise intervention (AE + RE) (Experimental): Physical exercise during neaodjuvant chemoradiation
  Interventions: Behavioral: combined aerobic exercise + resistance exercise intervention (AE + RE)
- Aerobic exercise prior to daily radiotherapy sessions (ExPR) (Experimental): Physical exercise during neaodjuvant chemoradiation
  Interventions: Behavioral: Aerobic exercise prior to daily radiotherapy sessions (ExPR)
- Usual care control (UC) (No Intervention): The control group will receive usual care and will be requested to maintain their usual daily physical activities.

INTERVENTIONS:
Behavioral: combined aerobic exercise + resistance exercise intervention (AE + RE) — The AE + RE intervention group will be offered a supervised exercise program which includes both aerobic and resistance exercise. Exercise sessions will take place twice a week with a duration of 60 minutes. The training load will be tailored to a patient's individual fitness level throughout the intervention. Patient will be asked to be physically active on an additional day in the week on their own (for at least 30 minutes at moderate intensity) according to the ACSM guidelines for patients with cancer.
  Arms: combined aerobic exercise + resistance exercise intervention (AE + RE)
Behavioral: Aerobic exercise prior to daily radiotherapy sessions (ExPR) — Patients in the ExPR in-hospital exercise intervention group will be offered an aerobic exercise program at moderate intensity. The exercise sessions will take place 5 days a week (only weekdays), and will have a duration of 30 minutes including a warming-up (5 min) and cooling-down (5 min). Total exercise volume will be aimed at 150 min per week. The sessions will take place within an hour before the daily radiotherapy session.
  Arms: Aerobic exercise prior to daily radiotherapy sessions (ExPR)

SUMMARY:
The goals of this study is to 1) evaluate feasibility and fidelity of a three-arm RCT containing a twice-weekly exercise intervention supervised by a first-line (oncology) physiotherapist and a 5-day weekly in-hospital exercise intervention versus usual care in patients with rectal cancer or esophageal cancer receiving NCRT, and 2) generate preliminary data on the variability in exercise responses on immune function, immune infiltration, and vascularisation of the tumour.

Participants will be randomized in one of three study arms: 1) AE + RE - group; combined moderate-to-high intensity aerobic exercise (AE) and resistance exercise (RE) twice a week supervised by a specially trained first-line physiotherapist, and a home-based moderate intensity aerobic exercise session once a week; 2) ExPR - group; in-hospital exercise intervention consisting of 30 min moderate intensity aerobic exercise within one hour prior to every radiotherapy session (five times a week); and 3) UC - group; a control group that receives usual care.

The main study parameters will be the feasibility in terms of trial participation rate and attendance, and intervention fidelity (e.g. extend of and reasons for adaptations to the exercise intervention). The secondary study parameters are the average effect sizes and measures of variability on immune function, infiltration and vascularisation. Measurements will take place at baseline, directly after finishing NCRT, and within a week before surgery.

DETAILED DESCRIPTION:
Strong evidence from randomized controlled trials (RCT) showed that physical exercise during chemotherapy or radiotherapy benefits physical fitness, muscle mass, muscle strength, fatigue, and health-related quality of life (HRQoL). Additionally, exercise may counteract treatment-related side effects and help prevent treatment modifications, which might improve survival. To date, the majority of RCTs examining the effects of exercise during cancer treatment have been conducted in patients with breast cancer or prostate cancer who were treated with curative intent. Due to differences in treatment trajectories and side effects, generalisability of these findings to patients with other types of cancer is limited. Additionally, widespread implementation of exercise in clinical cancer care is hampered by the lack of knowledge of the exercise effects on clinical outcome, e.g. tumour recurrence, progression and cancer-specific survival. Also, the causality and underlying physiological and biological mechanisms linking exercise to clinical outcome are largely unknown. This knowledge is essential to understand the potential and limitations of exercise as integral part of cancer care and to further optimize exercise interventions. Pre-clinical studies have shown that exercise can directly impact tumour growth and function as sensitizer for anticancer treatment. However, it is unclear whether these results can be translated to patients.

Standard treatment for patients with esophageal cancer and for a part of the patients with rectal cancer includes neoadjuvant chemoradiation treatment (NCRT), followed by a 6 - 12 weeks or 8 - 10 weeks waiting period prior to surgical resection, respectively. NCRT might reduce tumour size and even induce a pathological complete response. However, pathological complete response rate after NCRT is relatively low for these patient populations: 15-20% for rectal cancer and 30% for esophageal cancer. A part of patients with rectal cancer are treated with radiotherapy (50 Gray in 25 fractions of 2 Gray) for five weeks combined with the oral chemotherapy capecitabine. NCRT for patients with esophageal cancer includes radiotherapy (41.4 Gray in 23 fractions for 5 days a week) combined with the intravenous chemotherapies paclitaxel and carboplatin once a week for 5 weeks. Besides the curative value of NCRT it may cause severe treatment-related side effects including diarrhoea, fatigue, haematological toxicity, and neuropathy. Exercise training may counteract side effects such as fatigue, neutropenia, neuropathy, and gastrointestinal problems (e.g. nausea) while simultaneously improving physical fitness and HRQoL. Exercise frequency, intensity, timing and type may impact the effects of the intervention. For example, aerobic exercise at higher intensities may provide larger cardiovascular benefits, but may result in more gastrointestinal side effects. Therefore, it is important to study whether exercise is feasible during neoadjuvant chemoradiation, and whether exercise frequency, intensity, and timing can induce different effects. Thus, more knowledge is needed on the feasibility and effectivity of exercise prescriptions in patients with rectal or esophageal cancer, and the robustness of the potential exercise-induced effects across patient populations. Improving neoadjuvant treatment in these patients populations might enable more organ saving surgeries, and increase survival rates.

Potential mechanisms of exercise training influencing clinical and pathological response In addition to the well-established influence of physical exercise on physical fitness and the HRQoL in patients with cancer, pre-clinical studies showed that exercise training can directly influence tumour growth. To illustrate, studies in rodents revealed a few possible mechanisms by which exercise training can influence tumour physiology, including exercise-induced immune reactions, and alterations in vascularisation and perfusion of the tumour. Studies in mice showed exercise-induced immune reactions, stimulated by the release of epinephrine and the cytokine interleukin-6 (IL-6). IL-6 and epinephrine can initiate an immune response which mobilises, activates and redistributes natural killer (NK) cells. These processes have shown to stimulate the infiltration of activated NK cells in the tumour and to reduce tumour growth. Secondly, in mouse-models, exercise training showed to induce a 'normalisation' of the intratumoural vasculature, reducing hypoxia and thereby improving the chemotherapeutic and radiotherapeutic efficiency. Both pathways might contribute to a more rapid tumour regression. Due to differences between animal models and humans, including feasible exercise levels, tumour characteristics, metabolic rates and potential comorbidities, it is unclear whether these results can directly be translated to (wo)men.

The number of studies in patients investigating mechanistic pathways of exercise-induced tumour changes are scarce. Long-term exercise training as well as acute exercise bouts are characterised by specific physiological responses leading to immediate and chronic adaptations. Exploratory studies on exercise during neoadjuvant chemotherapy in patients provided initial support for the hypothesis that exercise can modulate several host- and tumour related pathways. These studies showed that exercise influenced circulating systemic factors, such as vascular endothelial growth factor (VEGF), Tumour Necrosis factor (TNF)-α, interleukins (ILs), and intracellular adhesion molecule (ICAM)-1. Due to the exercise-induced release of circulating systemic anti-inflammatory cytokines and angiogenic factors, aerobic training might improve immune activation in patients. Indeed, studies investigating the immune system showed that acute exercise induces a mobilisation of NK cells (and an improved NK-cell cytotoxicity in patients with cancer. In addition, data from our METRIC pilot trial in 14 patients with breast or colon cancer, showed that a 9-week exercise intervention during chemotherapy preserved NK-cell functionality (degranulation and cytotoxicity) compared to a reduction in the usual care control group, with a 10% difference between groups.

To our knowledge there are only two clinical trials in patients who investigated the influence of exercise training on tumour perfusion and vascularisation. In the study of Jones et al. among women with breast cancer, only limited data was available for perfusion assessments due to the relatively high proportion of patients with pathological complete responses. The study of Florez Bedoya et al. in patients with pancreatic cancer showed an increased number of vessels, elongated vessels, open vessels and an increased microvascular density in the tumour of patients who received an exercise intervention compared to historic control samples. Studies assessing changes in immune activation in the blood as well as intra-tumoural vascularisation and immune infiltration after exercise training during NCRT are non-existent in patients with rectal or esophageal cancer.

Another potential mechanism through which exercise may affect tumour response to NCRT in patients with rectal cancer is an altered microbiome. At the pathology department of Radboudumc, dr. Boleij and Prof. dr. Nagtegaal examine the mucosal and fecal microbiome in relation to colorectal cancer development and disease progression using in situ detection techniques and feces collections at multiple timepoints during disease trajectories. Exercise may have a positive effect on the microbiome, by modifying the microbiota and increases health-beneficial gut bacteria populations. An insight in changes in the microbiome after an exercise intervention during NCRT might provide valuable information about the tumour micro-environment. Hence, in this pilot study we want to exploratively include the collection of feces in patients with rectal cancer.

Besides the effects of exercise training after multiple sessions, pre-clinical studies showed that the induced effects of one exercise bout might already interfere with mechanisms underlying cancer progression and treatment response. Potential mechanisms for this acute phenomenon include mild hyperthermia, augmented tumour perfusion, reduced tumour hypoxia, and enhanced immune mobilisation. Even after one exercise bout these mechanisms may enhance tumour oxygenation and immunity, which could potentially, driven by accumulative effects of repeated acute exercise, result in improved radiotherapy efficacy.

An acute bout of exercise in healthy participants induces a large transient increase in peripheral blood lymphocyte counts, including NK cells and CD8+ T cells. In addition, an acute exercise bout can increase NK-cell cytotoxicity with 50 - 100%. Lymphocyte numbers return to below pre-exercise values 1-2 hours after exercise, possibly reflecting a redistribution of immune cells to peripheral tissue, which could be beneficial for immune surveillance. It was shown that acute exercise in healthy individuals selectively mobilises memory CD8+ T cells. Notably, Goedegebuure et al. showed that esophageal cancer patients enriched with circulating CD8+ memory T cells prior to the start of treatment were more likely to have a pathological complete response after NCRT. Also, high levels of CD8+ memory T cell infiltration in the tumour are associated with a good prognosis in both esophageal and colorectal cancer.

Besides the immune activation, pre-clinical studies showed that acute exercise might impact the tumour perfusion and hypoxia. As reported above, several pre-clinical studies report more patent and perfused vessels after exercise training, resulting in a larger and more homogeneously perfused tumour area. An acute reduction in hypoxia might make the tumour more sensitive to the radiotherapy. In addition, exercise-induced hyperthermia of the human body might induce vasodilatation, increase perfusion and make the tumour more permissible for immune cells. Consequently, linking the immune effects and perfusion effects of acute exercise to radiotherapy efficacy reveals the possibility of acute exercise as radiosensitizer. A close timing of an exercise session directly prior a radiotherapy session might be beneficial for the radiotherapy response. Exercise prior to a radiotherapy session was proven to be feasible and safe in patients with non-small cell lung carcinoma.

The feasibility and safety of an exercise intervention during NCRT in patients with rectal cancer and esophageal cancer has been evaluated in previous studies. High adherence rates and no adverse events related to the exercise intervention were reported in these studies, and most reported barriers were willingness to participate and recruitment of patients. We foresee that close collaborations with our multidisciplinary research team (e.g. clinical researchers, clinicians,specially trained physiotherapists, tumour immunologist, pathologist) and alignment of measurements with routine clinical practice will reduce these barriers. These previous studies explored the effects of exercise interventions during neoadjuvant therapy on physical activity, fitness, HRQoL, and post-operative complications. Additionally, exploratory studies detected that exercise during NCRT in patients with rectal cancer and esophageal cancer might lead to an augmented tumour regression. However, both in patients with rectal and esophageal cancer, there is only one RCT investigating the feasibility of a supervised exercise intervention during NCRT, and none of the currently performed studies included investigations of underlying mechanisms of action.

To our knowledge there is only one RCT evaluating the feasibility of aerobic exercise prior to each radiotherapy session during concomitant chemoradiotherapy (24). This small trial in patients with locally advanced non-small cell lung cancer showed that pre-radiotherapy exercise was safe and feasible.

We aim to conduct a three-arm pilot RCT in patients with rectal or esophageal cancer, while simultaneously collecting data on the underlying mechanisms through which exercise can influence tumour microenvironment. This pilot will investigate the feasibility of 1) AE + RT; an exercise intervention consisting of two exercise sessions per week combining moderate-to-high aerobic exercise (AE) and resistance exercise (RE) supervised by a first-line specially educated physiotherapist, and one home-based moderate intensity aerobic exercise session per week, 2) ExPR; in-hospital exercise intervention consisting of 30 min moderate intensity aerobic exercise sessions within one hour prior to every radiotherapy session (five times a week). Both interventions are similar in terms of weekly exercise volume. Simultaneously, this pilot will gather preliminary data on measures of variability on the potential efficacy of exercise on immune function, immune infiltration and vascularisation of both exercise interventions. Additionally, we will evaluate the acute immune response of one exercise session in patients in the ExPR group.

Knowledge on the feasibility and preliminary results of the underlying mechanisms of exercise regimes will be a first step towards improved supportive care for patients with rectal and esophageal cancer receiving neoadjuvant chemoradiation. If the preliminary results on underlying mechanisms are promising, we aim to write a grant application to set up a sufficiently powered multi-centre randomized controlled trial in cooperation with other large medical centres (e.g. Erasmus MC, Amsterdam UMC), focusing on the effects of exercise on tumour responses and underlying mechanisms.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with rectal or esophageal cancer
* Patients with rectal or esophageal cancer need to be scheduled for treatment with neoadjuvant chemoradiation therapy

  * Oral capecitabine combined with concurrent radiotherapy (50 Gy in 25 fractions) for rectal cancer
  * CROSS regimen (carboplatin, paclitaxel with concurrent 41.4 Gy in 23 fractions radiation) for esophageal cancer
* Aged > 18 years
* Provided written informed-consent

Exclusion Criteria:

* Unable to perform basic activities of daily living such as walking or biking
* Presence of other disabling co-morbidity that might hamper or endanger physical exercise e.g. heart failure, chronic obstructive pulmonary disease, orthopaedic conditions and neurological disorders
* Presence of cognitive disorders or severe emotional instability (e.g., Schizophrenia, Alzheimer, alcohol addiction)
* Immunodeficiency (primary or secondary)
* Insufficient mastery of the Dutch language
* Participation in another exercise and/or dietary intervention study at the same time.
* Already participating in structured vigorous aerobic and/or resistance exercise ≥ 2 times per week comparable to our intervention and planning to continue this throughout the period of neoadjuvant chemoradiation.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
Participation rate | 5 weeks (During intervention period)
  Participation will be assessed by calculating a rate between eligible patients and participating patients. An accrual rate lower than 20% will be defined as not feasible
Exercise intervention attendance | 5 weeks (During intervention period)
  Attendance will be assessed dividing the number of attended sessions by the number of prescribed sessions. The information will be collected using questionnaires and exercise-logs registered by the physical therapists (AE+RT arm) and researcher (ExPR arm). These logs will be collected by the researcher.
Intervention fidelity in terms of compliance | 5 weeks (During intervention period)
  Exercise intervention fidelity will be explored for both patient groups. Compliance will be evaluated by the session attendance.
Exercise relative dose intensity (ExRDI) | 5 weeks (During intervention period)
  ExRDI will be determined as the ratio of total completed to total planned cumulative exercises dose, expressed as a percentage.

SECONDARY OUTCOMES:
Body composition | 12-18 weeks (Baseline, post-intervention, pre-surgery)
  Measured by Body impedance analysis (BIA).
Estimated aerobic fitness | 12-18 weeks (Baseline, post-intervention, pre-surgery)
  Measured by Ästrand-Rhyming test in ml/kg/min
Muscle strength | 12-18 weeks (Baseline, post-intervention, pre-surgery)
  Estimated in kg by an indirect 1 RM legpress protocol.
Physical activity | 12-18 weeks (Baseline, post-intervention, pre-surgery)
  Measured by SQUASH (MET-score)
Health-related quality of life | 12-18 weeks (Baseline, post-intervention, pre-surgery)
  Measured by SF-36, PRO-CTCAE
Treatment toxicity | 12-18 weeks (Baseline, post-intervention, pre-surgery)
  Measured by PRO-CTCAE
Satisfaction | 12-18 weeks (Baseline, post-intervention, pre-surgery)
  Measured by a custom questionnaire
Immune cell function | 12-18 weeks (Baseline, post-intervention, pre-surgery)
  Measured by venous blood sampling and functional tests.
Immune cell mobilisation | 12-18 weeks (Baseline, post-intervention, pre-surgery)
  Measured by venous blood sampling and FACS
Immune cell infiltration | 12-18 weeks (Baseline, post-intervention, pre-surgery)
  Measured by immunohistochemistry of tumour tissue
Cytokines | 12-18 weeks (Baseline, post-intervention, pre-surgery)
  Measured by venous blood sampling
Tumour vascularisation | 12-18 weeks (Baseline, post-intervention, pre-surgery)
  Measured by immunohistochemistry of tumour tissue
Gut microbiome composition | 12-18 weeks (Baseline, post-intervention, pre-surgery)
  Measured by taxonomic features and alpha and beta diversity via 16S rRNA marker gene sequencing of feces samples

CONTACTS AND LOCATIONS:
Locations (1):
- Radboud Institute for Health Science, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided